CLINICAL TRIAL: NCT03362632
Title: A Prospective Study on Diagnosis and Treatment of End Stage Liver Disease Complicated With Infection (SESLDIP Study)
Brief Title: A Study on Diagnosis and Treatment of End Stage Liver Disease Complicated With Infection (SESLDIP Study)
Status: Unknown | Type: Observational
Last Known Status: Enrolling by invitation
Sponsor: Tongji Hospital (Other)
Responsible Party: Principal Investigator, Qin Ning, Director of Department of Infectious Disease, Tongji Hospital
Other Study IDs: SESLDIP study
Record Dates: First submitted 2017-11-22; First posted 2017-12-05 (Actual); Last update posted 2018-09-13 (Actual); Status verified 2017-11

CONDITIONS: End Stage Liver Disease; Infection; Spontaneous Bacterial Peritonitis
MeSH Terms: conditions — End Stage Liver Disease; Infections | interventions — Anti-Bacterial Agents

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Infection Group: Patients with end stage liver disease with SBP
  Interventions: Drug: Antibiotics
- Non-infection Group: Patients with end stage liver disease without SBP

INTERVENTIONS:
Drug: Antibiotics — This is an observation study, no specific antibiotics will be indicated during treatment.
  Groups: Infection Group

SUMMARY:
Spontaneous bacterial peritonitis (SBP) is a common complication of end-stage liver disease due to various causes. The initial anti-infective medication is appropriate and the patient's survival rate is closely related. Ascitic fluid bacterial culture takes a long time, the positive rate is low, it is difficult to guide the timely use of antimicrobial drugs, empirical medicine based on evidence-based medicine for SBP in patients with end-stage liver disease is essential. The American College of Hepatology and the European Society of Hepatology recommend the use of third-generation cephalosporins as the first choice of empirical therapy in patients with end-stage liver disease associated with community-acquired SBP. Patients with merger of hospital-acquired SBP with piperacillin / tazobactam or carbapenem +/- glycopeptide antibiotics is the first choice for empirical medication. There is no clear recommendation in China. In recent years, the conclusions of international clinical research in this area have been in disagreement with the recommendations. As a key factor in the selection of empirical antibiotics is local bacterial resistance data, these findings are difficult to evidence-based medicine for Chinese doctors. This project intends to observe the efficacy of different initial anti-infective regimens in Chinese patients with end-stage liver disease with SBP and 30-day and 60-day non-liver transplant survival rates, providing evidence-based medical evidence for the empirical use of such patients.

ELIGIBILITY:
Inclusion Criteria:

1. Meet the end-stage liver disease part of the type of standard (including slow plus acute liver failure, chronic liver failure, cirrhosis decompensation);
2. age> 18 years old
3. ascites nucleated cell count> 250 × 106 / L;
4. Unable to obtain ascites specimens or ascites nucleated cells count does not meet the conditions of 3) are required abdominal examination tenderness (+), rebound tenderness (+), abdominal ultrasound can detect ascites, and procalcitonin (PCT) > 0.5ng / ml, hs-CRP> 10ng / ml

Exclusion Criteria:

1. history of abdominal surgery within 4 weeks;
2. secondary peritonitis;
3. tuberculous peritonitis;
4. Malignant tumor;
5. patients who use hormones or immunosuppressants;
6. AIDS patients;
7. heart failure or respiratory failure;
8. merge other parts of the infection;
9. died within 48h;
10. liver transplantation during observation;
11. Diagnosis of spontaneous bacterial peritonitis is the use of carbapenems or third-generation cephalosporins / enzyme inhibitors, piperacillin / enzyme inhibitor antibiotics

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Patients with chronic liver disease
Sampling Method: Non-Probability Sample
Enrollment: 400 (Estimated)
Dates: Start 2018-07-01 (Actual); Primary Completion 2018-12-31 (Estimated); Study Completion 2019-06-30 (Estimated)

PRIMARY OUTCOMES:
Complete response rate to empirical antibiotic treatment | 6 months
  The percentage of patients who achieved complete recovery from combined infection after empirical antibiotic treatment

SECONDARY OUTCOMES:
Non-liver transplant survival | 6 months
  Non-liver transplant survival rate at 30 days, 60 days and 6 months after empirical antibiotic treatment
Hospitalization time | 6 months
  Days of hospitalization after empirical antibiotic treatment

CONTACTS AND LOCATIONS:
Locations (1):
- Department of Infectious Disease, Tongji Hospital, Tongji Medical College, Huazhong University of Science and Technology, Wuhan, Hubei, China

IPD SHARING:
Plan to Share IPD: Undecided